CLINICAL TRIAL: NCT01024881
Title: Influence of the Shoulder Position on the Catheter Tip Location During Infraclavicular Subclavian Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jae-Hyon Bahk, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHBahk_CVC shoulder position
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Catheter Tip Location
Keywords: catheterization success rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Active Comparator): neutral shoulder position during infraclavicular subclavian catheterization
  Interventions: Procedure: neutral shoulder position
- group 2 (Experimental): lowered shoulder position during infraclavicular subclavian catheterization
  Interventions: Procedure: lowered shoulder position

INTERVENTIONS:
Procedure: neutral shoulder position — neutral shoulder position during infraclavicular subclavian catheterization
  Arms: group 1
Procedure: lowered shoulder position — lowered shoulder position during infraclavicular subclavian catheterization
  Arms: group 2

SUMMARY:
Infraclavicular approach of the subclavian veins is commonly used for central venous access. Aberrant locations of catheter tip are frequently quoted for this approach, but few studies have been performed to document the relationship between the shoulder position and catheter tip location. This prospective study was performed to assess the influence of the shoulder position on the safe and proper placement of infraclavicular subclavian catheters.

ELIGIBILITY:
Inclusion Criteria:

* adult patients requiring central venous catheterization due to major procedures such as neurosurgery or thoracic surgery.

Exclusion Criteria:

* chest deformities,
* coagulopathy,
* diaphragmatic dysfunction,
* pulmonary malformation,
* history of prior clavicle fracture, or
* infection over the puncture site.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2008-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
location of the catheter tip | at the end of surgery

SECONDARY OUTCOMES:
catheterization success rate | immediately after catheterization

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea